CLINICAL TRIAL: NCT03563092
Title: Closed Suction Drain vs no Drain on Symptomatic Seroma Formation After Laparoscopic Inguinal Hernia Repair
Acronym: SALHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMSALHS
Record Dates: First submitted 2018-05-28; First posted 2018-06-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Inguinal Hernia Without Obstruction or Gangrene
Keywords: Complete Inguinal Hernia; Inguinoscrotal Hernia; Laparoscopic hernia repair
MeSH Terms: conditions — Gangrene | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Open-label, randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lap Inguinal Hernia repair with Drain (Experimental): A (14 French sizes) closed suction drain will be placed in preperitoneal space after laparoscopic inguinal hernia (TEP/TAPP) surgery.
  Interventions: Procedure: Laparoscopic Inguinal Hernia (TEP/TAPP) Surgery
- Lap Inguinal Hernia repair without Drain (Active Comparator): No drain will be placed after laparoscopic inguinal hernia (TEP/TAPP) surgery.
  Interventions: Procedure: Laparoscopic Inguinal Hernia (TEP/TAPP) Surgery

INTERVENTIONS:
Procedure: Laparoscopic Inguinal Hernia (TEP/TAPP) Surgery — Standardized minimally invasive approach to inguinal hernia repair

SUMMARY:
The current study aims to determine whether a use of closed suction drain following laparoscopic inguinal hernia surgery performed for an inguinoscrotal variety can decrease the incidence of symptomatic seroma formation requiring interventions and thus, prevent postoperative morbidity.

DETAILED DESCRIPTION:
Patients with laparoscopic inguinal repair, TEP as well as TAPP approach, which matches the inclusion criteria will be randomized intraoperatively, based on a complete assessment of eligibility, just before the mesh placement.

Patients recruited in closed suction drain arm will receive suction drain(14 French sizes) in preperitoneal space via a separate incision. The patients without drain arm, the regular postoperative course will be followed.

The drain will be removed once the output falls below 50 ml per day. Both groups will be followed up until three months post-surgery.

Clinical suspicion of seroma in symptomatic patients will be confirmed by ultrasound. Seroma will be managed conservatively till three weeks in the post-op period.

ELIGIBILITY:
Inclusion Criteria:

All patients having an inguinoscrotal hernia (complete type)

Exclusion Criteria:

Obstructed, incarcerated or strangulated hernia Patients unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients developing symptomatic seroma requiring intervention after surgery | Month 3
  The patients developing symptomatic seroma after hernia surgery, assessed by clinical and radiological evaluation, which needs intervention in form of needle aspiration or sac excision.

SECONDARY OUTCOMES:
Surgical site infection | Month 3
Postoperative Pain | Day 1
  Measured by Visual Analogue Pain Scale
Recurrence | Month 3
  Early recurrence of Hernia

OTHER OUTCOMES:
Factors affecting seroma | Day 7
  To study the various factors associated with seroma like patients demographics, surgeon related factors, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chinnusamy Palanivelu, MS,MCh,FRCS,FACS, Study Chair — Gem Hospital and Research Center, Coimbatore, India; Sandeep C. Sabnis, MS,DNB, Principal Investigator — Gem Hospital and research center, Coimbatore, India
Locations (1):
- Sandeep C. Sabnis, Coimbatore, Tamil Nadu, India